CLINICAL TRIAL: NCT03934944
Title: A Feasibility Study to Compare Usual Methods of Patient Education With a Multi-media Presentation and Weekly 'Foot-alerts' Using 21st Century Technologies to Improve Patient Diabetic Foot Care Knowledge and Practices
Brief Title: A Feasibility Study Comparing Usual Foot Education and Phone App Alerts in Patients With Increased Risk of Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: Kuwait Foundation for the Advancement of Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RA HM-2018_044
Record Dates: First submitted 2019-03-06; First posted 2019-05-02 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer
Keywords: Patient education; Prevention; Smart phone application
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone application arm (Experimental): Participants will have access to a educational video and foot alerts at weekly intervals to supplement usual Podiatry care and education.
  Interventions: Device: Phone application
- Usual care (Other): Participants will have Podiatry care and education.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Phone application — Weekly foot alerts and educational video
  Other Names: MyU smart phone application
  Arms: Phone application arm
Other: Usual care — Usual routine of diabetic foot education
  Other Names: Routine Podiatry education
  Arms: Usual care

SUMMARY:
The purpose of this study is to compare foot care knowledge, behaviour and glycaemic control in patients at increased risk of diabetic foot ulcers. Participants will receive either usual diabetic foot care education and follow-up as per evidence-based guidelines or usual care and follow-up, supplemented with an educational video and weekly foot alerts via a phone application.

DETAILED DESCRIPTION:
It is recommended that patients who are at moderate or high risk of diabetic foot ulcer (DFU) are seen by a healthcare professional for foot review every 2-6 months. Yet, diabetic foot ulcers remain the leading cause of non-traumatic lower limb amputation with an amputation occurring every 20 secs. This suggests that additional information and prompts, as well as regular follow-up, are required. Additionally, long term diabetic foot complications including loss of protective pain sensation are related to poor glycaemic control.

This single blinded randomised study aims to determine if weekly foot alerts (a total of 12 alerts cycled over 12-months), delivered by the MyU phone application in combination with usual education routes and follow-up, improves patient foot care behaviour and foot care knowledge. Using standardized questionnaires at baseline and 12-months. Furthermore, does the frequency of viewing/engaging in foot alert content influence foot care knowledge and behaviour.

Secondary objectives are to determine: 1) if individuals who receive 7-foot review appointments in a 12-month period have better foot care knowledge and behaviour when compared to those seen less frequently regardless of educational route. 2) Baseline and 12-months HbA1c blood test will be measured to establish if any changes occurred between the two groups.

Expected results: The investigators hypothesized that participants randomised to the intervention group (Phone app) will have improved foot care knowledge and foot health behaviours.

Sample size: 100 patients with a 1:1 ratio

Quality Assurance:

A standard operating procedure based on established diabetic foot screening tools will be used to ensure the inter-rater reliability of foot assessment.

Educational material will go through back translation to ensure the accuracy of the content. Feedback on content, meaning and usability of the English and Arabic documents from a sample of 10 participants will be sought.

To maintain investigator blinding the participants will be escorted to the video viewing room by a research coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 21 yrs or
* Type 2 Diabetes Mellitus or Type 1 Diabetes Mellitus greater than 5-yrs
* At least one diabetic foot risk factor (i.e Loss of Pain Sensation Peripheral Arterial Disease etc)
* Ability to understand Arabic or English to a skill listening level 3 and speaking level +2 (Interagency Language Roundtable).
* Own a smartphone and access to the internet
* The ability to understand the study procedures and to comply with them for the entire length of the study
* Resident in Kuwait

Exclusion Criteria:

* Chronic kidney disease stage 3 or above
* Cognitive impairment
* Acute psychiatric illness
* Hearing or visual impairment that would mean the intervention would not be understood
* phone application inaccessible for more than 4 continuous weeks
* Refusal to give written informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in foot care knowledge as measured by the adapted foot care knowledge test | 12 months
  Change in the adapted Diabetic Foot Care Knowledge test (Pollock et al. 2004 and Rheeder et al. 2008) score between baseline and 12-months in the two groups This 12-question test has a maximum score of 12, and a minimum score of 0. Each correct answer is given one point, where a low score denotes low knowledge and high score denotes high knowledge. For each group a mean will be calculated and significance of differences will be tested using the students two tailed unpaired T-Test.
Change in foot care behaviour as measured by the SDSCA | 12 months
  SDCS questionnaire includes a number of domains which evaluate different aspects of patient behaviour performed during the previous week. Each domain has one or more questions that are marked between 0-7. The domains are:
  1. Foot care: total of 9 questions with maximum score 9x7 = 63, the greater the score the better the behaviour
  2. Diabetes Management: 4 questions in diabetes management, maximum score 4x7 = 28, the greater the score the better the behaviour
  3. Smoking habits: number of cigarettes per day, the greater the number the worse the behaviour
  These measures allow formulation of a composite reflection in changes in the patient's behaviour between baseline and 12-months in the two groups. Differences will be tested using the students two-tailed unpaired T-Test.

SECONDARY OUTCOMES:
Change in HbA1c from baseline | 12 months
  Change in HbA1c measurement taken from venous blood supply at baseline and 12-months between intervention and control group.
Proportion of participants who developed a new diabetic foot ulcer | 12 months
  Case report form. Diabetic foot ulcer is defined as a wound below the ankle in someone with diabetes and will be classified using the University of Texas Wound classification System.

CONTACTS AND LOCATIONS:
Overall Officials: Kay Scarsbrook Khan, BSc, Principal Investigator — Dasman Diabetes Institute; Ebaa Al Ozairi, MD, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No